CLINICAL TRIAL: NCT02452879
Title: The Effectiveness, Superiority and Safety of EA on OAB:Multi-center Randomized Controlled Trial
Brief Title: Treatment, Parallel Assignment, Double Blind (Subject, Outcomes Assessor), Efficacy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Capital Medical University (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Baohui Jia, Deputy director of Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z121107001012148
Record Dates: First submitted 2015-05-02; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Electroacupuncture; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electroacupuncture group (Experimental): Needle on bilateral BL33 acupoint 50-60mm with a 60°angle. A feeling of soreness and distension will be felt when needling into the 3rd posterior sacral foramina(S3). Needle with 75mm long needle. An electric stimulator is put on. SDZ-V electric stimulator (produced by Suzhou Medical Instrument Co.Ltd). continuous wave(CW), 10Hz. Stop turning up the current intensity when patients could not stand. 3 times a week. Once every other day. The treatment period lasts eight weeks. totally 24 times.30min/time.
  Interventions: Device: Electroacupuncture
- Placebo group (Placebo Comparator): with the patient in the prone position. The acupoint routine disinfection of skin, and then the fixed pad is adhered on the acupoint. The 1.5 inches blunt tip needle pierce through the fixed pad, then it reaches the surface of the skin, uniform lifting thrusting and twirling all 3 times but do not pierce the skin. Then connect the electric acupuncture apparatus with special power supply wire electrode (special power line as the middle wire cut, looks as normal; that electroacupuncture instrument display connected to the state, but the actual without electricity), in the bilateral Zhongliao points, Hui Yang points on the needle handle; the period of treatment and the other manipulation of the placebo group are same as the deep needling acupoint group.
  Interventions: Device: Sham Electroacupuncture
- Solifenacin Succinate group (Active Comparator): Solifenacin Succinate Tablets (made by the Anse Tailai Pharmaceutical (China) R & D limited company) 5mg, 1 tablets each time, 1 times / day, oral administration of 30min before meal, even for 8 weeks.
  Interventions: Drug: Solifenacin Succinate

INTERVENTIONS:
Device: Electroacupuncture — For the deep needling acupoint group, needle on bilateral BL33 50-60mm with a 60°angle. A feeling of soreness and distension will be felt when needling into the 3rd posterior sacral foramina(S3). Needle with 75mm long needle. An electric stimulator is put on. SDZ-V Hua Tuo Brand electric stimulator (produced by Suzhou Medical Instrument Co.Ltd). continuous wave(CW), 10Hz. Stop turning up the current intensity when patients could not stand. 3 times a week. Once every other day The treatment period lasts eight weeks. totally 24 times.30min/time.
  Arms: Electroacupuncture group
Device: Sham Electroacupuncture — with the patient in the prone position. The acupoint routine disinfection of skin, and then the fixed pad is adhered on the acupoint. The 1.5 inches blunt tip needle pierce through the fixed pad, then it reaches the surface of the skin, uniform lifting thrusting and twirling all 3 times but do not pierce the skin. Then connect the electric acupuncture apparatus with special power supply wire electrode (special power line as the middle wire cut, looks as normal; that electroacupuncture instrument display connected to the state, but the actual without electricity), in the bilateral Zhongliao points, Hui Yang points on the needle handle; the period of treatment and the other manipulation of the placebo group are same as the deep needling acupoint group.
  Arms: Placebo group
Drug: Solifenacin Succinate — made by the Anse Tailai Pharmaceutical (China) R & D limited company) 5mg / tablet
  Arms: Solifenacin Succinate group

SUMMARY:
The purpose of this study is to determine whether electroacupuncture is effective in the treatment of overactive bladder.

DETAILED DESCRIPTION:
Patient registry: Participants experiencing overactive bladder will be recruited from hospital outpatients and clinic-community. the diagnosis was made by the urologists. the random number table was generated by the Computer.

Sample size: According to the preliminary experiment combined the literature. Sample size is based on the primary outcome. The first step: one-tailed test: the electroacupuncture group vs Solifenacin group is 79.5% VS 54.8%( α=0.05, β=0.20, n=51). The second step: two-tailed test :the electroacupuncture group vs Placebo group is 54.5% VS 20.9%,(α=0.05, β=0.20, n=37). To combine the first and second step, 51 cases in each group are needed. Allowing for a 10% dropout, 57 cases in each group are needed. So we set the sample size is 60.

Quality control

1. Strict training on staff participating in the trial.
2. Rigorous control of the process of randomization.
3. Specific inclusion and exclusion criteria.
4. Strict outcome assessors and statisticians.
5. The standard of the drugs, acupuncture apparatus, inspection equipment are consistant.
6. Outcome assessment, completion of case report forms and data management will be under strict supervision.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of overactive bladder.
2. Frequent micturition.（average urinary frequency of ≥8 voids per day）
3. No relevant drug use within 2 weeks and no acupuncture treatment within 1 month before the study; not in other clinical trials.
4. Self-reported bladder symptoms ≥3 months
5. Capable of giving informed consent .
6. Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Frequent micturition and urinary urgency are secondary to other diseases.
* Clinical diagnosis of simple stress urinary incontinence.
* Patients with urinary track infection and vagenal infection.
* Patients with implantable pelvic stimulator.
* Current use of electric therapy on pelvic area/back/legs.
* Current use of clostridium botulinum therapy on vesical or pelvic muscles.
* participation in any clinical inverstigation involving or impacting gynecological/urinary/renal function.
* Suffering from severe cardiac/hepatic/renal injury or cognitive disorder/aphasia/ dysphrenia/malnutrition, or in poor perform status and unable to cooperate.
* Patients in gestation and in lactation period.
* Patients in coagulation disorders or taking anticoagulation drugs.
* People with cardiac pacemaker or metal allergy.
* Patients having got eletroacupunture therapy or solifenacin in 4 weeks before the study.
* Patients are afraid of needles.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean frequency of micturitions per 24 hours | 4, 8 weeks in treatment, 12th and 24th weeks of follow-up
  Mean daily micturition frequency = Sum of 3-day micturition frequency in a week/3 . The investigator gets the frequency of mictuitions by micturition diary.Mean daily micturition frequency will be calculated based on the micturition diary at week 0(baseline), 2, 4, 6, 8, 20, 32.

SECONDARY OUTCOMES:
The response rate of improvement in symptoms | 8 weeks in treatment, The average response rate of improvement in global response during 8 weeks in treatment. The response rate in first 4 weeks in treatment, 12 and 24 weeks of follow-up will also be evaluated
  GRA（Global response assessments）will be used to grade:
  The overall response will be assessed by patient self-rating scale. There are seven levels which will be graded by patients based on their situation: significant deterioration, moderate deterioration, mild deterioration, no change, mild improvement, moderate improvement, significant improvement in symptoms (compared with their condition before treatment). The moderate and significant improvement will be defined as effective treatment while others will be defined as ineffective ones according to the patients' options. The response rate will be calculated separately.
  Response rate= Effective number of patients in each group/ Total number of patients in each group×100%

OTHER OUTCOMES:
Patient-Rated Global Assessments of treatment Benefit, Satisfaction, and Willingness to Continue (The BSW) | Week 4th , 8th in treatment , 12nd and 24th of follow-up
  For therapeutic benefit scores, treatment will be regarded beneficial if scores are above (3). The patient-Rated global assessment of treatment benefit will be calculated according to scores of patients in each group.
  For treatment satisfaction scores, scores above (3) will be recorded as satisfaction. Treatment satisfaction scores will be calculated based on scores of patients in each group.
  The willing to continue the treatment scores, scores above (3) will be recorded as willing to continue the treatment scores, the scores will be calculated based on the scores of patients in each group.
The mean number of daily urgency micturition, nocturia, leakage of urine, the mean degree of daily urgency micturition | 4 weeks, 8 weeks in treatment, 12nd and 24th weeks of follow-up.
  mean degree of daily urgency micturition will be captured at week 0(baseline), 2, 4, 6, 8, 20, 32 based on the micturition diary.
Daily mean incidence of urgency micturition (%), daily mean incidence of leakage of urine(%) | Week 0(baseline), 4, 8, 12 and 24 of follow-up
  Daily mean incidence of urgency micturition and leakage of urine will be calculated. Urgency incontinence, stress incontinence and unconscious leakage of urine will be included.
  Incidence of urgency micturition (%):the frequency of urgency micturition in a week based on three day urine diary/ three days' total times of urination in ×100% Incidence of leakage of urine (%): the frequency of leakage of urine in a week based on three day bladder diary/ three days' total times of urination ×100%
Oab-Q | on Friday of week 0 (baseline), 4, 8, 12, 24
  The patients will be asked to write the questionnaires which have a total of 33 questions. The degree of which the patients suffer from overactive bladder including urgency micturition, pollakiuria , nocturia, urge incontinence will be assessed by the first 8 questions. 1-6 points will be given for each question and all the points will be added and converted to 0-100 points which suggest higher severity with higher scores. The effect of symptoms on life will be assessed by the rest questions which will be divided to disease problems, sociality, mood, sleeping. The points of each part which includes 2-5 questions will be added separately as subscale scores. All of them will be added and converted to 0-100 points which will be the score for quality of life representing better quality with higher points.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Baohui, Master, Study Chair — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Hargreaves E, Baker K, Barry G, Harding C, Zhang Y, Kandala NB, Zhang X, Kernohan A, Clarkson CE. Acupuncture for treating overactive bladder in adults. Cochrane Database Syst Rev. 2022 Sep 23;9(9):CD013519. doi: 10.1002/14651858.CD013519.pub2. PMID 36148895